CLINICAL TRIAL: NCT04334031
Title: Deployment o the Multidisciplinary Prospective Cohort Imminent
Acronym: IMMINeNT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: FHU IMMINeNT (Unknown); FHU PRECISE: Projet Fédératif Hospitalo-Universitaire PREcision health in Complex Immune-mediated inflammatory diseaSEs (Unknown); Fond de dotation de la Société Française de Dermatologie (SFD) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018_82; 2019-A01309-48 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-03-10; First posted 2020-04-03 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Chronic Inflammatory Disease; Angioedema; Severe Asthma; Lupus; Atopic Dermatitis; Psoriatic Arthritis; Multiple Sclerosis; Systemic Sclerosis; Behçet Disease
Keywords: Immune Mediated Inflammatory Diseases (IMIDs); biomarker; cohort study; quality of life; disease severity
MeSH Terms: conditions — Angioedema; Asthma; Dermatitis, Atopic; Arthritis, Psoriatic; Multiple Sclerosis; Scleroderma, Systemic; Behcet Syndrome | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMMINeNT cohort (Experimental)
  Interventions: Genetic: Biobanking with genetic analysis; Other: SF-12 questionnaire

INTERVENTIONS:
Genetic: Biobanking with genetic analysis — Patients included in the IMMINeNT cohort will be collected 7 blood samples for the research project at each revaluation visit. For patients who accepted, genetic analysis (DNA analysis) will be done on a part of those samples.
Other: SF-12 questionnaire — Patients included in the IMMINeNT cohort will be asked to complete SF-12 quality of life questionnaire.

SUMMARY:
Immune-mediated inflammatory diseases (IMIDs) most often affect young patients and have high impact on morbidity and mortality with a significant alteration in the quality of life of patients with professional, social and emotional repercussions.

Beyond this burden, IMIDs share many common pathophysiological mechanisms and treatments, known as "targeted therapies". Despite progress in this field, much remains to be done in clinical, therapeutic and fundamental research to address the efficacy, resistance and side-effects of treatment.

These similarities between IMIDs have led the FHU IMMINeNT to propose the creation of a prospective, multidisciplinary clinical-biological database (IMMINeNT cohort), associated to a biobank, of patients with IMIDs. The main objectives of this database will be to identify new prognostic and therapeutic biomarkers in order to develop new therapeutic targets and biomarkers, to identify prognostic factors and determinants related to the activity, severity and quality of life of patients with IMIDs as well as to the response and tolerance to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient followed for their IMID in one of the departments of the Lille University Hospital participating in the study (dermatology, internal medicine, neurology, pneumology and rheumatology)
* Social insured
* Have the capacity to understand the study requirements, provide written informed consent, and comply with the study data collection procedures.

Exclusion Criteria:

* Administrative reasons: inability to receive informed information, inability to participate in the entire study, lack of coverage by the social security system.
* Pregnant or breastfeeding woman
* Persons deprived of liberty
* Protected minors or adults
* Persons who have refused or are incapable of giving informed consent
* Persons in Emergency Situations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Change of SLEDAI for lupus | once a year for 10 years
  for lupus:Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) The SLEDAI score calculator consists of a list of 24 items, 16 clinical and 8 laboratory results.The total score falls between 0 and 105, with higher scores representing increased disease activity.
Change of Medsger score | once a year for 10 years
  Medsger Score estimates disease involvement of each organ (heart, vessels, skin, brain, kidney, gut, muscle, joint and loss of weight,) ranging from 0 to 4 (0: normal, 1: mild, 2: moderate, 3: severe, 4: terminal). The score ranges from 0 to 36 points.A higher score means a worse outcome.
Change of EDSS for multiple sclerosis | once a year for 10 years
  for multiple sclerosis:Expanded Disability Status Scale (EDSS) The EDSS quantifies disability in eight Functional Systems (FS) by assigning a Functional System Score (FSS) in each of these functional systems EDSS steps 1.0 to 4.5 refer to people with MS who are fully ambulatory. EDSS steps 5.0 to 9.5 are defined by the impairment to ambulation.EDSS score is a specific multiple sclerosis scale, from 0 (normal neurological status) to 10 (death kinked to sclerosis).
Change of BASDAI for psoriatic arthristis | once a year for 10 years
  For psoriatic arthritis:Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) he BASDAI consists of a 0 - 10 scale measuring discomfort, pain, and fatigue (0 being no problem and 10 being the worst problem) in response to six questions asked of the patient pertaining to the five major symptoms of AS: Fatigue/Spinal pain/Arthralgia (joint pain) or swelling/Enthesitis, or inflammation of tendons and ligaments (areas of localized tenderness where connective tissues insert into bone)/Morning stiffness duration/Morning stiffness severity.
Change of Longhurst criteria for hereditary angioedema | once a year for 10 years
  for hereditary angioedema: Longhurst criteria
Change of number of flares for atopic dermatitis | once a year for 10 years
  There is no validated score for atopic dermatitis and severe asthma.For atopic dermatitis, disease activity will be assessed by the number of flares per month with any affected body surface area (ACS) and the number of flares with body surface area >20%.
Change of number of exacerbations for severe asthma | once a year for 10 years
  For severe asthma, disease activity will be assessed by the number of exacerbations per month, where an exacerbation is defined as a loss of control resulting in an increase in beta2mimetic intake (>2 times daily compared to usual) and/or asthma-related limitation of daily activity and/or peak-flow change >30% from baseline on at least 2 consecutive days)
Change of 12-Item Short-Form Health Survey (SF-12) - quality of life scale | once a year for 10 years
  Health-related Quality of Life variable measured using the Short Form Health Survey (SF12): 12-item self-report that assesses physical and mental health related quality of life. Results are expressed in terms of two meta-scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The PCS and MCS scores have a range of 0 to 100 and were designed to have a mean score of 50. Higher scores indicate better physical functioning.
number of participant with severe infectious events | once a year for 10 years

CONTACTS AND LOCATIONS:
Overall Officials: David Launay, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France